CLINICAL TRIAL: NCT00737828
Title: A Randomised Controlled Trial of the Utility of Cardiopulmonary Exercise (CPX) Testing for Preoperative Risk Stratification to Guide Perioperative Care and Thereby Reduce Postoperative Morbidity
Brief Title: Cardiopulmonary Exercise Testing and Preoperative Risk Stratification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mike Grocott, Professor, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07/0114; 07/H0716/55 (Other: NHNN REC Number); PB-PG-0906-11426 (Other Grant/Funding Number: UK National Institute of Health Research (NIHR))
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer; Anaesthesia; Critical Illness
Keywords: Cardiopulmonary exercise test; CPX; CPEX; surgical outcome; colorectal surgery; risk stratification
MeSH Terms: conditions — Colorectal Neoplasms; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Control - Standard Perioperative Pathway, clinician decides post-operative care environment (usual care)
  Interventions: Other: Perioperative care pathway guided by CPX results
- B (Experimental): Intervention - Perioperative care pathway guided by CPX Results i.e.anaerobic threshold & ventilatory equivalents
  Interventions: Other: Perioperative care pathway guided by CPX results

INTERVENTIONS:
Other: Perioperative care pathway guided by CPX results — * AT > 11ml/min/kg no myocardial ischaemia or Ve/VO2 <35 - Level 1 Ward Care
  * AT > 11ml/min/kg with myocardial ischaemia or Ve/VO2 >35 - Level 2/3 (ITU) Critical Care Unit
  * AT <11mls/min/kg - Level 2/3 Critical Care Unit
  * AT <8mls/min/kg - Level 2/3 Critical Care Unit/ consider cancellation or alternative procedure

SUMMARY:
The investigators would like to evaluate the use of cardiopulmonary exercise tests (CPX) in guiding the care pathway of patients undergoing colorectal operations. In the intervention group care will be guided by CPX results and in the control group care will be guided by the doctors assessment. The investigators would like to assess the impact of this on patient outcome, patient satisfaction and resource usage.

DETAILED DESCRIPTION:
Each year 20000 UK patients die within 30 days of surgery. It seems that in the UK a patient's chances of becoming seriously unwell or dying following surgery is higher than in comparable countries. Fewer beds in the UK are given over to Intensive Care than in these other countries. Closer attention to the care given after operations, which can be achieved on intensive care units (ICU), almost certainly reduces the chances of serious illness following major surgery. An increase in the number of intensive care unit beds in the UK is extremely unlikely. Better use of the available intensive care beds could be achieved by allocating them where they are believed to improve outcome (following surgery) and by allocating them to patients most likely to benefit.

Tests used to assess risk of surgery to patients are largely ineffective. Cardiopulmonary exercise tests (CPX) seem to be effective at identifying patients at risk of death or serious illness post surgery. This information has been used in studies to select patients for ICU beds and reduce deaths. The studies so far have limitations in their design and scope which means we can't be certain this approach works in the UK.

We suggest a study to answer this question more conclusively and more specifically in UK patients. We will randomly divide patients between two groups. In the 1st group choice of postoperative care environment is based on best current practice and in the other group we will make these decisions (critical care or ward) based on the results of the CPX.

We hope that the benefits will include less patients becoming seriously ill or dying and shorter stays in hospital after surgery following major operations. We also hope the information will help patients understand the risks of their operation better and therefore make better informed decisions. This may also reduce the overall cost of surgery for hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years age
2. Males
3. Females
4. Listed for elective(non-emergency) colorectal surgery

Exclusion Criteria:

1. Age < 18 years age
2. Patient unwilling/unable to consent
3. Adults with learning disabilities or dementia
4. Prisoners
5. Any contraindication to cardiopulmonary exercise testing (as outlined by *American Association of Anaesthesia:

   * Acute MI (3-5 days)
   * Unstable angina
   * Uncontrolled arrhythmias
   * Syncope
   * Acute endocarditis
   * Acute myocarditis
   * Acute pericarditis
   * Symptomatic severe aortic stenosis
   * Uncontrolled heart failure
   * Acute pulmonary embolism or infarction
   * Thrombosis of lower extremities
   * Dissecting aneurysm
   * Uncontrolled asthma
   * Pulmonary oedema
   * Room air desaturation at rest <85%
   * Respiratory failure
   * Acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise Mental impairment leading to inability to co-operate
6. Patients already enrolled in an interventional study
7. Previous CPX test result recorded in the medical notes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity (presence or absence of POMS defined morbidity) | Day 5

SECONDARY OUTCOMES:
Post operative morbidity domains e.g. gastrointestinal, renal, pulmonary | Day 5
Total postoperative ITU bed utilisation | End of hospital stay i.e. day of hospital discharge
Total postoperative bed utilisation | End of hospital stay i.e. day of hospital discharge
ITU re-admission | End of hospital stay i.e. day of hospital discharge
Death | Should death occur
SF36 (compared with SF36 at baseline) | 12 months post day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael PW Grocott, Study Director — University College, London; Paula Meale, Principal Investigator — University College, London; Michael Mythen, Principal Investigator — University College, London; Ayo Oshowo, Principal Investigator — Whittington Hospital NHS Trust; Mervyn Singer, Principal Investigator — University College, London; Geoff Bellingan, Principal Investigator — University College London Hospitals; Kay Mitchell, Principal Investigator — University College, London; Hasan Muktar, Principal Investigator — The Whittington Hospital Hospital NHS Trust; Alistair Windsor, Principal Investigator — University College London Hospitals; Jim Down, Principal Investigator — University College London Hospitals; Martin B Kuper, Principal Investigator — Whittington Hospital NHS Trust; Denny ZH Levett, Principal Investigator — University College, London; Phil Hennis, PhD, Principal Investigator — UCL; Alasdair O'Doherty, MSc, Principal Investigator — UCL; Alec Engledow, Principal Investigator — UCLH; Aundrea Mulreany, Principal Investigator — Whittington Hospital; Carolyn Dr Way, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Karen Linford, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Clare Bolger, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Paul Nichols, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Kim Golder, Principal Investigator — University Hospital Southampton NHS Foundation Trust; John S Knight, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Michael Celinski, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Grace Adesina, Principal Investigator — University College London Hospitals
Locations (3):
- United Kingdom (3):
  - Whittington Hospital NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Southampton University Hospitals NHS Trust, Southampton